CLINICAL TRIAL: NCT00155168
Title: Quantitative Analysis of SMN1 and SMN2 Gene Based on DHPLC System: Establishing a Novel Highly Efficient and Reliable SMA Carrier Screening Test
Brief Title: Quantitative Analysis of SMN1 and SMN2 Gene Based on DHPLC System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361700452
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2004-04

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal muscular atrophy (SMA); SMN1/SMN2 gene; denaturing high-performance liquid chromatography (DHPLC); multiplex PCR; gene dose; carrier test
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
In this project, we will establish the efficient and accurate gene dose determination system by combining the heterodulex analysis and gene dose analysis on DHPLC platform based on various quantitative and multiplex PCR strategies and applying on detecting the carriers- in- risk and patients with spinal muscular atrophy.This method is, therefore, based on the observation that the amount of PCR product generated from each site of amplification is proportional to the amount of starting template. Detection of PCR products is carried out on DHPLC, which provide the sensitivity required for the detection of the single-copy dosage changes.

DETAILED DESCRIPTION:
Proximal spinal muscular atrophy is an autosomal recessive disorder with an overall incidence of 1 in 10000 live births and a carrier frequency of 1 in 50. This severe neuromuscular disease is characterized by a degeneration and loss of alpha motor neurons of the spinal cord anterior horn cells, which results in progressive symmetrical weakness, atrophy of the proximal voluntary muscles, and infant death.

Two most identical copies of SMN gene, telomeric SMN (SMN1) and centromeric SMN (SMN2), have been identified. These two SMN genes are highly homologous and differing in only five nucleotide exchanges within their 3' regions. These variations do not alter the encoded amino acids. These nucleotide differences located in exons 7 and 8, allow SMN1 gene to be distinguished from SMN2 gene.

It has been reported that more than 95% of SMA patients were homozygous deletion of SMN1 gene. Therefore, the detection of the absence of SMN1 can be a useful tool for SMA diagnosis. Furthermore, because of the high incidence of SMA, the high carrier frequency of at least 1 in 50, the severity of the disease in the patients, and the lack of effective of treatment, carrier testing for SMN1 deletion is an important question in genetic counseling. However, a highly homologous SMN2 gene also exits and hampers the detection of the loss of SMN1 which makes the detection of SMA carrier test difficult.

Here, we present a new, rapid, simple and high reliable method to detect the SMN1 deletion and to determine the copy number of the SMN1 and SMN2 by denaturing high-performance liquid chromatography (DHPLC). DHPLC is a novel, simple, fast and non gel-base method that is very sensitive and specific for detection DNA variations. Furthermore, we describe a multiplex PCR strategy to determine the SMN1 and SMN2 genes copy number in order to avoid bias due to fluctuations in the copy number of SMN genes. The assay uses the X-linked CYBB gene and KRIT1 gene as standards to determine the relative gene dosage of SMN1 and SMN2 genes. We demonstrate that this assay is able to accurately distinguish 2 gene copies from 4 gene copies and it can identify SMA carriers and normal populations by the accurate determination of SMN copy number.

This project will contribute to apply this novel, fast, and reliable tool for diagnosis of SMA and carrier detection of SMN1 and SMN2 genes by using DHPLC system.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Spinal muscular atrophy

Exclusion Criteria:

* nil

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500
Dates: Start 2004-04

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ning su, MD,PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- Dept of Medical Genetics;National Taiwan University Hospital, Taipei, Taiwan